CLINICAL TRIAL: NCT05591469
Title: Respiratory Measurement Using Infrared Camera and Electrical Impedance Tomography for Sedation in Patients Undergoing TURP/TURB Under Spinal Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 4-2022-0864
Record Dates: First submitted 2022-10-13; First posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Patients Undergoing Transurethral Prostate or Cystectomy Under Spinal Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Noncontact Respiration monitoring group (Experimental)
  Interventions: Device: IR Camera
- Contact Respiration monitoring group (Experimental)
  Interventions: Device: Electrical Impedance Tomography

INTERVENTIONS:
Device: IR Camera — the respiration parameters are measured using an IR camera.
  Arms: Noncontact Respiration monitoring group
Device: Electrical Impedance Tomography — the respiration parameters are measured using an electrical impedance tomograhy.
  Arms: Contact Respiration monitoring group

SUMMARY:
Tidal volume may be the most important technical indicator for ventilation. Measuring tidal volume can be used as an indicator of how effective a patient's gas exchange is, and can also be used as a predictive indicator to indirectly predict the severity of respiratory disease. This tidal volume can be measured using spirometry and pneumotachograph, and the lung function of the patient can be assessed directly or indirectly through the respiratory volume and air flow velocity. In addition, the measurement itself can change the patient's breathing pattern, and for accurate measurement, it has to be carried out in a certain space, so there is a limitation in that it is difficult to measure in a hospital bed or in a laboratory. To overcome this limitation, various methods have been introduced. The basic principle is that the tidal volume is directly proportional to the movement of the chest and proportional to the change in the length of the circumference of the chest. Over the past decade, several studies have been conducted to measure respiratory mechanics in a non-invasive way. Methods using thoracic impedance, acoustic monitoring, strain gauges, and magnetometers have been developed. Non-invasive, non-contact imaging methods have also been developed, such as thermal image, structured light plethysmography (SLP), and optoelectronic plethysmography (OEP). Therefore, in this study, the thoracic movement due to respiration was measured with a non-invasive method (IR camera), and the accuracy was compared through the impedance change obtained through impedance tomography to evaluate the effectiveness of the non-invasive equipment.

ELIGIBILITY:
Inclusion Criteria:

* A male aged 19 years or older
* normal BMI
* patients undergoing transurethral prostate or cystectomy under spinal anesthesia

Exclusion Criteria:

* Presenting alteration in respiratory function detected by functional analysis of lung volume and capacity- pneumonectomy patient, severe ipsilateral destroyed lung patient
* Inability to understand or perform the procedure.
* ASA class 4, 5

Ages: 19 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
The accuracy of respiration measurements | Experiment period about 20 minutes
  The accuracy respiration measurements between IR camera and electrical impedance tomography.

CONTACTS AND LOCATIONS:
Overall Officials: Jeongmin Kim, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kim J, Kwon JH, Kim E, Yoo SK, Shin CS. Respiratory measurement using infrared thermography and respiratory volume monitor during sedation in patients undergoing endoscopic urologic procedures under spinal anesthesia. J Clin Monit Comput. 2019 Aug;33(4):647-656. doi: 10.1007/s10877-018-0214-4. Epub 2018 Nov 14. PMID 30426322
- [Background] Kwon J, Kwon O, Oh K, Kim J, Shin CS, Yoo SK. Thermodiluted relative tidal volume estimation using a thermal camera in operating room under spinal anesthesia. Biomed Eng Online. 2022 Sep 7;21(1):64. doi: 10.1186/s12938-022-01028-0. PMID 36071495